CLINICAL TRIAL: NCT06254209
Title: Randomized and Double-blind Study to Evaluate the Physiological Effects on the Skin of 3 Food Supplements Versus Placebo in 40-60 Years Old Female Subjects
Brief Title: Study to Evaluate the Physiological Effects on the Skin of 3 Food Supplements Versus Placebo in 40-60 Years Old Female Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nexira (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: COS04
Record Dates: First submitted 2023-12-18; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo
- Verum1 (Experimental): Combination of clove (Syzygium aromaticum) and immortelle (Helichrysum italicum) extracts
  Interventions: Dietary Supplement: Botanicals extracts
- Verum2 (Experimental): Olive fruit extract (Olea europaea)
  Interventions: Dietary Supplement: Botanicals extracts
- Verum3 (Experimental): Hibiscus flower extract (Hibiscus sabdariffa)
  Interventions: Dietary Supplement: Botanicals extracts

INTERVENTIONS:
Dietary Supplement: Botanicals extracts — Powder included in capsules for daily administration
  Arms: Verum1; Verum2; Verum3
Dietary Supplement: Placebo — Maltodextrin included in capsules for daily administration
  Arms: Placebo

SUMMARY:
The objective is to evaluate the effects on the skin of 3 foods supplements compared to placebo after daily intake for 3 months in female subjects presenting healthy skin.

Skin parameters measured are: the firmness of the skin and other biomechanical skin properties (elasticity, tonicity, density), cellulitis visibility, radiance complexion, skin condition (microrelief, skin barrier function and moisturizing)

DETAILED DESCRIPTION:
Study design: Monocentric, randomized, double blind, placebo controlled, 3 groups in parallel.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Phototype II to IV (Fitzpatrick)
* Visual skin radiance score (face) ≤ 7 (0 to 9 points numeric scale)
* Tactile skin firmness score (cheek) ≤ 7 (0 to 9 points numeric scale)
* Visual cellulite score (thigh) ≥ 3 (0 to 9 points numeric scale)

Exclusion Criteria:

* Chronic pathology or systemic disorder
* Subjects presenting imperfections on the test sites
* Pregnant or who are planning to become pregnant
* Medication or condition that may interfere with tested outcomes

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Firmness of the skin | Day 0 (inclusion) and Day 84 (last visit)
  Cutometry measurements using Cutometer (cheekbone)

SECONDARY OUTCOMES:
Skin elasticity and tonicity | Day 0 (inclusion) and Day 84 (last visit)
  Cutometry measurements using the Cutometer (cheekbone)
Skin density | Day 0 (inclusion) and Day 84 (last visit)
  Ultrasound imaging device (lower cheek)
Score of fine lines visibility on face, assessed by panelist (trained technician) | Day 0 (inclusion) and Day 84 (last visit)
  10 points numeric scale: 0 (not visible) to 9 (highly visible)
Score of skin radiance of face, assessed by panelist (trained technician) | Day 0 (inclusion) and Day 84 (last visit)
  10 points numeric scale: 0 (dull) to 9 (radiant)
Score of nourishing aspect (hydration and quality aspect) of face, assessed by panelist (trained technician) | Day 0 (inclusion) and Day 84 (last visit)
  10 points numeric scale: 0 (malnourished) to 9 (nourished)
Score of skin firmness (tactile pinch of right cheek), assessed by panelist (trained technician) | Day 0 (inclusion) and Day 84 (last visit)
  10 points numeric scale: 0 (sagging) to 9 (firm)
Score of skin softness (tactile perception of right cheek), assessed by panelist (trained technician) | Day 0 (inclusion) and Day 84 (last visit)
  10 points numeric scale: 0 (rough) to 9 (soft)
Score of cellulite visibility (right thigh), assessed by panelist (trained technician) | Day 0 (inclusion) and Day 84 (last visit)
  10 points numeric scale: 0 (not visible) to 9 (highly visible)
Dimpled skin - volume (mm3) of humps and dimples | Day 0 (inclusion) and Day 84 (last visit)
  Picture acquisition by fringe projection (on tight) and software integration
Dimpled skin - surface (mm2) of humps and dimples | Day 0 (inclusion) and Day 84 (last visit)
  Picture acquisition by fringe projection (on tight) and software integration
Skin luminosity - CIELAB (L*a*b) | Day 0 (inclusion) and Day 84 (last visit)
  Standardized pictures acquisitions (face) and software integration
Skin color texture - Haralick parameter (contrast & entropy - no unit) | Day 0 (inclusion) and Day 84 (last visit)
  Standardized pictures acquisitions (face) and software integration
Skin specular reflectance (spectral reflectance - no unit) | Day 0 (inclusion) and Day 84 (last visit)
  Standardized pictures acquisitions (face) and software integration
Skin roughness (mean height - µm) | Day 0 (inclusion) and Day 84 (last visit)
  Standardized 3D pictures acquisitions (cheek) and software integration
Skin barrier function (g/h/m²) | Day 0 (inclusion) and Day 84 (last visit)
  Trans-epidermal water loss (forearm)
Skin moisture (%) | Day 0 (inclusion) and Day 84 (last visit)
  Reflected electromagnetic probe (forearm)
Self perceived questionnaire (4 scales) | Day 0 (inclusion), Day 42 (intermediate) and Day 84 (last visit)
  Questionnaire (Satisfied, Somewhat satisfied, Somewhat unsatisfied, Unsatisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Intertek, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided